CLINICAL TRIAL: NCT00572442
Title: Magnetocardiography (MCG) in Asymptomatic Individuals - Pilot Trial
Status: Withdrawn | Type: Observational
Why Stopped: sponsor funding
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: CardioMag Imaging (Industry)
Responsible Party: Kirsten Tolstrup, MD, Cedars-Sinai Medical Center
Other Study IDs: 13939
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Non-invasive heart scan; MCG; Cardiac Risk Factors; healthy volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Subjects without any cardiovascular risk factors:
  1. Age ≥ 45 in men; Age ≥ 55 in women.
  2. Hypertension: BP > 140/90 mmHg or on BP meds.
  3. Diabetes Mellitus: Known fasting blood sugar >126 mg/dl or on DM meds.
  4. Dyslipidemia: On lipid lowering medication or LDL ≥ 160 mg/dl in absence of other risk factors; ≥ 130 mg/dl if other non-diabetic risk factors; ≥ 100 mg/dl if diabetic. Known HDL < 40 mg/dl.
  5. Cigarette smoking (past or present).
  6. Family history of premature CAD in first degree relatives: Age < 55 in men; Age < 65 in women.
- 2: Subjects with 1 cardiovascular risk factor (listed above)
- 3: Subjects with 2 cardiovascular risk factors (listed above)
- 4: Subjects with more than 2 cardiovascular risk factors (listed above)

SUMMARY:
The purpose of this research study is to perform serial magnetocardiographs (MCG)and cardiovascular risk factor assessments on individuals with no symptoms or history of heart disease. This small sized study of MCG in healthy individuals will allow for data collection for power analysis for a larger prospective trial.

Volunteers are not compensated or paid.

DETAILED DESCRIPTION:
The Magnetocardiography (MCG) has been approved by the U.S Food and Drug Administration (FDA) as a tool to measure the heart's magnetic field.However, it is not yet approved for the specific diagnosis of coronary artery disease.

The MCG scan is entirely non-invasive, rapid and no risk, since it does not require stress provocation, radiation, or use of medication or contrast.

In this study, the MCG will be used to compare the scans of normal, healthy volunteers to those which have been previously or are currently being collected in subjects with known heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without chest pain and known heart diseases.
* Subjects > or = 18 years of age.

Exclusion Criteria:

* Heart disease patients
* Patients with chest pain
* Subjects with magnetic metal fragments in the head or torso
* Subjects unable to consent
* Minors < 18 years of age
* Subjects unable to lie flat for the examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: individuals without symptoms or history of heart disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Tolstrup, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States